CLINICAL TRIAL: NCT05033691
Title: A Multi-center, Open-label, Randomized, Two-arm Study, to Evaluate the Efficacy of Osimertinib With Early Intervention SRS Treatment Compared to the Continuation of Osimertinib Alone, in Patients With EGFR Mutated NSCLC and Asymptomatic Brain Metastases.
Brief Title: A Study to Evaluate the Efficacy of Osimertinib With Early Intervention SRS Treatment Compared to the Continuation of Osimertinib Alone, in Patients With EGFR Mutated NSCLC and Asymptomatic Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, MEIRROVITZ AMICHAY, Principle investigator, oncologist and radiation specialist, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUNG-OSIME-SRS
Record Dates: First submitted 2021-07-04; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: NSCLC; EGFR Gene Mutation; EGF-R Positive Non-Small Cell Lung Cancer; Non-small Cell Lung Cancer; Brain Metastases
Keywords: nsclc; non-small cell lung cancer; EGFR Gene Mutation; EGF-R Positive Non-Small Cell Lung Cancer; EGFR; Brain Metastases; osimertinib; tagrisso; SRS; stereotactic radiosurgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Early SRS treatment with SoC (Experimental): Stereotactic surgery (SRS) to the brain metastases and continuation of Osimertinib, at 2 month (8 weeks) post Osimertinib start
  Interventions: Radiation: Stereotactic surgery
- SoC Tagrisso treatment only (Active Comparator): continuation of osimertinib alone
  Interventions: Radiation: Stereotactic surgery

INTERVENTIONS:
Radiation: Stereotactic surgery — At two month (8 weeks) post Osimertinib start, patients will be randomized into one of the two study arms. Arm A patients will be treated with stereotactic surgery (SRS). In both arms Osimertinib treatment will continue.

SUMMARY:
This study involves patients with EGFR-mutated NSCLC and asymptomatic brain metastases. This is an open-label, randomized study, comparing the continuation of Osimertinib treatment alone to Osimertinib treatment combined with early intervention stereotactic radiosurgery (SRS). The current first line of care for EGFR-mutated NSCLC is administration of Osimertinib, a small molecule that penetrates the blood brain barrier (BBB) well and controls majority, but not all, of the brain metastases. We hypothesize that relatively early intervention with SRS to brain metastases that are still visualized by MRI 2 months-post initiation of Osimertinib treatment, LUNG- will improve long term brain control, cognitive abilities and potentially overall survival. Patients with EGFR-mutated NSCLC and asymptomatic brain metastases will be treated with Osimertinib for 2 months. Brain MRI scans will be collected pre-Osimertinib and 2 months after treatment start. Patients with asymptomatic brain metastases present after 2 months of Osimertinib will be randomized into one of two study arms. Arm A patients will be treated with SRS while continuing Osimertinib, while arm B patients will continue with Osimertinib alone. Patients will be assessed based on brain and whole body progression by RECIST. Patients will also be assessed for CNS-PFS and body-PFS, cognitive function, Quality of life and overall survival status via routine follow-up tests.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed metastatic NSCLC, not amenable to curative surgery or curative radiotherapy.
2. Documented EGFR mutation (at any time since the initial diagnosis of NSCLC) known to be sensitive to Osimertinib - These include exon 19 del; L858R (exon 21); G719X (exon 18); L861G (exon 21); S768I (exon 20) and T790M (exon 20) NOTE: Mutation analysis is to be done as per local practice.
3. An MRI showing brain metastases. At randomization, number of brain lesions is under 20. Patients with over 20 brain lesions at randomization MRI will be suitable for whole brain radiation, and will not be randomized.
4. Brain metastases are asymptomatic or with minor symptoms (ECOG≤2) at study randomization.
5. ECOG performance status ≤2 and a minimum life expectancy of at least 6 months
6. Must be eligible and receive Osimertinib as their anti EGFR TKI at time of randomization.
7. Must be eligible for SRS treatment at time of randomization.
8. Provided written informed consent.
9. Be male or female and at least 18 years of age on the day of signing informed consent.
10. Female patients:

    1. Willing to use adequate contraceptive measures until 6 weeks after the final dose of study treatment
    2. Not breast feeding
    3. Have a negative pregnancy test prior to the start of dosing if of childbearing potential or have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:
    4. Post-menopausal, defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments ii. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution iii. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
11. Male patients who are willing to use barrier contraception (i.e. condoms) until 4 months after the final dose of study treatment.

Exclusion Criteria:

* a. Prior treatment with:

  1. Anti EGFR TKI treatment.
  2. Checkpoint inhibitors immunotherapy for metastatic NSCLC.
  3. Whole brain radiation (WBRT) and/or Stereotactic Radiosurgery (SRS).
  4. Medications or herbal supplements known to be potent inducers of CYP3A4 and are unable to stop use within the recommended wash out period prior to receiving the first dose of Osimertinib.
  5. An investigational drug within five half-lives of the compound.
  6. Any other cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of entry to the study.

     b. Systemic progression under Osimertinib treatment between screen and randomization systemic scan, per RECIST1.1.

     c. Spinal cord compression unless asymptomatic and stable. d. Leptomeningeal disease. e. Moderate or severe symptomatic brain metastases defined as per Radiation Therapy Oncology Group acute morbidity grade 3 to 4.

     NOTE: Grade 3 refers to neurological findings requiring hospitalization for initial management. Grade 4 refers to serious neurological impairment including paralysis, coma or seizures more than three times per week despite medication and requires hospitalization.

     f. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.

     g. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Osimertinib.

     h. Involvement in the planning and conduct of the study i. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain control: CNS-PFS | Change in lesion size in the CNS will be followed and assessed at screen, Randomization, 2 month after Randomization, then every 3 month
  Lesions that did not disappear after two months of Osimertinib treatment will be better controlled with SRS

SECONDARY OUTCOMES:
whole body PFS | Change in lesion size in the whole body will be followed and assessed at screen, Randomization, 2 month after Randomization, then every 3 month
  Whole body progression will be delayed when Osimertinib is combined with early treatment of SRS
Cognitive function | Change in patient cognitive function will be followed and assessed at screen, Randomization, 2 month after Randomization, then every 3 month
  Patient cognitive function will improve after SRS treatment
Quality of life (QOL) | Change in patient quality of life will be followed and assessed at screen, Randomization, 2 month after Randomization, then every 3 month
  Patient QOL will improve after SRS treatment
Time to whole brain radiation | Status will be checked at every visit and follow up
  Time until whole brain radiation will be given will prolong for patients who receive early SRS treatment
Overall survival (OS) | Status will be checked at every visit and follow up
  Patient OS will improve after SRS treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Data for individual participants will be collected anonymously via the study CRF, data will be analyzed statistically and published.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Chen Z, Fillmore CM, Hammerman PS, Kim CF, Wong KK. Non-small-cell lung cancers: a heterogeneous set of diseases. Nat Rev Cancer. 2014 Aug;14(8):535-46. doi: 10.1038/nrc3775. PMID 25056707
- [Background] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929
- [Background] Yang JC, Wu YL, Schuler M, Sebastian M, Popat S, Yamamoto N, Zhou C, Hu CP, O'Byrne K, Feng J, Lu S, Huang Y, Geater SL, Lee KY, Tsai CM, Gorbunova V, Hirsh V, Bennouna J, Orlov S, Mok T, Boyer M, Su WC, Lee KH, Kato T, Massey D, Shahidi M, Zazulina V, Sequist LV. Afatinib versus cisplatin-based chemotherapy for EGFR mutation-positive lung adenocarcinoma (LUX-Lung 3 and LUX-Lung 6): analysis of overall survival data from two randomised, phase 3 trials. Lancet Oncol. 2015 Feb;16(2):141-51. doi: 10.1016/S1470-2045(14)71173-8. Epub 2015 Jan 12. PMID 25589191
- [Background] Teijeira S, Navarro C. [Dystrophinopathies: concept and diagnostic methodology]. Neurologia. 1994 May;9(5):191-7. No abstract available. Spanish. PMID 8024825
- [Background] Martinez P, Mak RH, Oxnard GR. Targeted Therapy as an Alternative to Whole-Brain Radiotherapy in EGFR-Mutant or ALK-Positive Non-Small-Cell Lung Cancer With Brain Metastases. JAMA Oncol. 2017 Sep 1;3(9):1274-1275. doi: 10.1001/jamaoncol.2017.1047. PMID 28520828
- [Background] Magnuson WJ, Lester-Coll NH, Wu AJ, Yang TJ, Lockney NA, Gerber NK, Beal K, Amini A, Patil T, Kavanagh BD, Camidge DR, Braunstein SE, Boreta LC, Balasubramanian SK, Ahluwalia MS, Rana NG, Attia A, Gettinger SN, Contessa JN, Yu JB, Chiang VL. Management of Brain Metastases in Tyrosine Kinase Inhibitor-Naive Epidermal Growth Factor Receptor-Mutant Non-Small-Cell Lung Cancer: A Retrospective Multi-Institutional Analysis. J Clin Oncol. 2017 Apr 1;35(10):1070-1077. doi: 10.1200/JCO.2016.69.7144. Epub 2017 Jan 23. PMID 28113019
- [Background] Duggirala KB, Lee Y, Lee K. Chronicles of EGFR Tyrosine Kinase Inhibitors: Targeting EGFR C797S Containing Triple Mutations. Biomol Ther (Seoul). 2022 Jan 1;30(1):19-27. doi: 10.4062/biomolther.2021.047. PMID 34074804
- [Background] Wang C, Lu X, Lyu Z, Bi N, Wang L. Comparison of up-front radiotherapy and TKI with TKI alone for NSCLC with brain metastases and EGFR mutation: A meta-analysis. Lung Cancer. 2018 Aug;122:94-99. doi: 10.1016/j.lungcan.2018.05.014. Epub 2018 May 18. PMID 30032853
- [Background] Wang J, Xia TY, Wang YJ, Li HQ, Li P, Wang JD, Chang DS, Liu LY, Di YP, Wang X, Wu WZ. Prospective study of epidermal growth factor receptor tyrosine kinase inhibitors concurrent with individualized radiotherapy for patients with locally advanced or metastatic non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e59-65. doi: 10.1016/j.ijrobp.2010.12.035. Epub 2011 Feb 23. PMID 21345607
- [Background] Du XJ, Pan SM, Lai SZ, Xu XN, Deng ML, Wang XH, Yao DC, Wu SX. Upfront Cranial Radiotherapy vs. EGFR Tyrosine Kinase Inhibitors Alone for the Treatment of Brain Metastases From Non-small-cell Lung Cancer: A Meta-Analysis of 1465 Patients. Front Oncol. 2018 Dec 12;8:603. doi: 10.3389/fonc.2018.00603. eCollection 2018. PMID 30619745
- [Background] Chang WS, Kim HY, Chang JW, Park YG, Chang JH. Analysis of radiosurgical results in patients with brain metastases according to the number of brain lesions: is stereotactic radiosurgery effective for multiple brain metastases? J Neurosurg. 2010 Dec;113 Suppl:73-8. doi: 10.3171/2010.8.GKS10994. PMID 21121789
- [Background] Mohammadi AM, Recinos PF, Barnett GH, Weil RJ, Vogelbaum MA, Chao ST, Suh JH, Marko NF, Elson P, Neyman G, Angelov L. Role of Gamma Knife surgery in patients with 5 or more brain metastases. J Neurosurg. 2012 Dec;117 Suppl:5-12. doi: 10.3171/2012.8.GKS12983. PMID 23205782
- [Background] Grandhi R, Kondziolka D, Panczykowski D, Monaco EA 3rd, Kano H, Niranjan A, Flickinger JC, Lunsford LD. Stereotactic radiosurgery using the Leksell Gamma Knife Perfexion unit in the management of patients with 10 or more brain metastases. J Neurosurg. 2012 Aug;117(2):237-45. doi: 10.3171/2012.4.JNS11870. Epub 2012 May 25. PMID 22631694
- [Background] Gerstenecker A, Nabors LB, Meneses K, Fiveash JB, Marson DC, Cutter G, Martin RC, Meyers CA, Triebel KL. Cognition in patients with newly diagnosed brain metastasis: profiles and implications. J Neurooncol. 2014 Oct;120(1):179-85. doi: 10.1007/s11060-014-1543-x. Epub 2014 Jul 18. PMID 25035099
- See also: Grambsch, P. M., & Therneau, T. M. (1994). Proportional hazards tests and diagnostics based on weighted residuals. Biometrika, 81(3), 515-526 — https://mayoclinic.pure.elsevier.com/en/publications/proportional-hazards-tests-and-diagnostics-based-on-weighted-resi